CLINICAL TRIAL: NCT01443858
Title: Meclizine as a Potential Smoking Cessation Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Philip Morris USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00030282
Record Dates: First submitted 2011-09-29; First posted 2011-09-30 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Cigarette Smoking; Meclizine; Nicotine Patch
MeSH Terms: conditions — Smoking Cessation; Cigarette Smoking | interventions — Meclizine; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo + Nicotine Patch (Active Comparator): Subjects in this group will take placebo meclizine daily for the three weeks prior to their quit date. Subjects will also apply a 21mg/24h nicotine patch daily starting in the second week of pre-quit treatment. Placebo meclizine will be administered in two doses each day.
  Interventions: Drug: Nicotine Patch; Drug: Placebo
- 25mg Meclizine + Nicotine Patch (Experimental): Subjects in this group will take 25mg of meclizine daily for the three weeks prior to their quit date. Subjects will also apply a 21mg/24h nicotine patch daily starting in the second week of pre-quit treatment. Meclizine will be administered in two doses each day.
  Interventions: Drug: Meclizine; Drug: Nicotine Patch
- 50mg Meclizine + Nicotine Patch (Experimental): Subjects in this group will take 50mg of meclizine daily for the three weeks prior to their quit date. Subjects will also apply a 21mg/24h nicotine patch daily starting in the second week of pre-quit treatment. Meclizine will be administered in two doses each day.
  Interventions: Drug: Meclizine; Drug: Nicotine Patch

INTERVENTIONS:
Drug: Meclizine — Pre-Quit Period: In this group, participants will take meclizine daily during the three week pre-quit period. The meclizine will be taken in two doses daily, one capsule with breakfast and one with dinner.
  Other Names: Antivert
  Arms: 25mg Meclizine + Nicotine Patch; 50mg Meclizine + Nicotine Patch
Drug: Nicotine Patch — Pre-Quit Period: During weeks two and three, participants will apply active 21mg/24h nicotine patches daily.
  Post-Quit Period: Following the quit-day these participants will apply active nicotine patches daily using the following dose schedule: 21mg/24h for four weeks, 14mg/24h for one week, and 7mg/24h for one week.
  Other Names: Nicoderm
Drug: Placebo — Pre-Quit Period: In this group, participants will take placebo capsules daily during the three week pre-quit period. The placebo will be taken in two doses daily, one capsule with breakfast and one with dinner.
  Arms: Placebo + Nicotine Patch

SUMMARY:
The purpose of this study is to evaluate whether meclizine, an antihistamine used to prevent or treat motion sickness, can help smokers quit smoking. This study will also investigate the potential relationship between genes you have inherited and success in quitting smoking.

ELIGIBILITY:
Inclusion Criteria:

* Have no known serious medical conditions;
* Are 18-65 years old;
* Smoke an average of at least 10 cigarettes per day;
* Have smoked at least one cumulative year;
* Have an afternoon expired air carbon monoxide (CO) reading of at least 10ppm;
* Express a desire to quit smoking in the next thirty days.
* Potential subjects must agree to use acceptable contraception during their participation in this study.

Potential subjects must agree to avoid the following during their participation in this study:

* participation in any other nicotine-related modification strategy outside of this protocol;
* use of tobacco products other than cigarettes, including pipe tobacco, cigars, e-cigarettes, snuff, and chewing tobacco;
* use of experimental (investigational) drugs or devices;
* use of illegal drugs;
* use of opiate medications
* use of anti-histamines;
* use of alcohol (during first three weeks of study participation).

Exclusion Criteria:

* Inability to attend all required experimental sessions;
* Hypertension (systolic >140 mm Hg, diastolic >100 mm Hg, coupled with a history of hypertension); subjects with no previous diagnosis of hypertension may have a screening blood pressure up to 160/100.
* Hypotension with symptoms (systolic <90 mm Hg, diastolic <60 mm Hg).
* Participants with a history of hypertension may, however, be allowed to participate in the study if the study physician or physician assistant determines that the condition is stable, controlled by medication, and in no way jeopardizes the individual's safety.
* Coronary heart disease;
* Lifetime history of heart attack;
* Cardiac rhythm disorder (irregular heart rhythm);
* Chest pains (unless history, exam, and ECG clearly indicate a non-cardiac source);
* Cardiac (heart) disorder (including but not limited to valvular heart disease, heart murmur, heart failure);
* History of skin allergy;
* Active skin disorder (e.g., psoriasis) within the last five years, except minor skin conditions (including but not limited to facial acne, minor localized infections, and superficial minor wounds);
* Liver or kidney disorder (except kidney stones, gallstones);
* Gastrointestinal problems or disease other than gastroesophageal reflux or heartburn;
* Active ulcers in the past 30 days;
* Currently symptomatic lung disorder/disease (including but not limited to chronic obstructive pulmonary disease (COPD), emphysema, and asthma);
* Brain abnormality (including but not limited to stroke, brain tumor, head injury and seizure disorder);
* Migraine headaches that occur more frequently than once per week;
* Recent, unexplained fainting spells;
* Problems giving blood samples;
* Diabetes treated with insulin; non-insulin treated diabetes (unless glucose is less than 180mg/dcl and HbA1c is less than 7%);
* Current cancer or treatment for cancer in the past six months (except basal or squamous cell skin cancer);
* Other major medical condition;
* Current psychiatric disease (with the exception of anxiety disorders, obsessive compulsive disorder (OCD) and ADHD);
* Current depression;
* Bulimia or anorexia;
* Pregnant or nursing;
* Smokes more than one cigar a month;
* Regular alcohol use;
* Significant adverse reaction to nicotine patches or meclizine in the past.
* Current participation or recent participation (in the past 30 days) in another smoking study at our center or another research facility.
* Current participation in another research study.

Use (within the past 30 days) of:

* Illegal drugs (or if the urine drug screen is positive),
* Experimental (investigational) drugs;
* Psychiatric medications including antidepressants, anti-psychotics or any other medications that are known to affect smoking cessation (e.g. clonidine);
* Smokeless tobacco (chewing tobacco, snuff), pipes or e-cigarettes;
* Wellbutrin, bupropion, Zyban, Chantix, varenicline, nicotine replacement therapy or any other smoking cessation aid.

Use (within the past 14 days) of:

* Opiate medications for pain or sleep (non-opiate medication for pain or sleep will be allowed);
* Benzodiazepines, antihistamines or other drugs with significant sedating or anticholinergic activity that may interact with meclizine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jed E Rose, Ph.D., Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Duke Center for Nicotine and Smoking Cessation Research, Charlotte, North Carolina
  - Duke Center for Nicotine and Smoking Cessation Research, Durham, North Carolina
  - Duke Center for Nicotine and Smoking Cessation Research, Raleigh, North Carolina
  - Duke Center for Nicotine and Smoking Cessation Research, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 9/16/11 and ended on 11/30/12. Of the 146 subjects consented during this period, 72 were in our Charlotte, NC office, 45 were in our Durham, NC office and 29 were in our Raleigh, NC office. Of the 146 subjects consented during this study only 75 subjects met all study criteria and were assigned to a study arm.
Groups:
- Control: Subjects in this group will take placebo meclizine daily for the three weeks prior to their quit date. Subjects will also apply a 21mg/24h nicotine patch daily starting in the second week of pre-quit treatment. Placebo meclizine will be administered in two doses each day.
  Nicotine patches: Pre-Quit Period: During weeks two and three, participants will apply active 21mg/24h nicotine patches daily.
  Post-Quit Period: Following the quit-day these participants will apply active nicotine patches daily using the following dose schedule: 21mg/24h for four weeks, 14mg/24h for one week, and 7mg/24h for one week.
- 25mg Meclizine: Subjects in this group will take 25mg of meclizine daily for the three weeks prior to their quit date. Subjects will also apply a 21mg/24h nicotine patch daily starting in the second week of pre-quit treatment. Meclizine will be administered in two doses each day.
  Meclizine: Pre-Quit Period: In this group, participants will take meclizine daily during the three week pre-quit period. The meclizine will be taken in two doses daily, one capsule with breakfast and one with dinner.
  Nicotine patches: Pre-Quit Period: During weeks two and three, participants will apply active 21mg/24h nicotine patches daily.
  Post-Quit Period: Following the quit-day these participants will apply active nicotine patches daily using the following dose schedule: 21mg/24h for four weeks, 14mg/24h for one week, and 7mg/24h for one week.
- 50mg Meclizine: Subjects in this group will take 50mg of meclizine daily for the three weeks prior to their quit date. Subjects will also apply a 21mg/24h nicotine patch daily starting in the second week of pre-quit treatment. Meclizine will be administered in two doses each day.
  Meclizine: Pre-Quit Period: In this group, participants will take meclizine daily during the three week pre-quit period. The meclizine will be taken in two doses daily, one capsule with breakfast and one with dinner.
  Nicotine patches: Pre-Quit Period: During weeks two and three, participants will apply active 21mg/24h nicotine patches daily.
  Post-Quit Period: Following the quit-day these participants will apply active nicotine patches daily using the following dose schedule: 21mg/24h for four weeks, 14mg/24h for one week, and 7mg/24h for one week.
Period: Overall Study
Arm/Group | Control | 25mg Meclizine | 50mg Meclizine
Started | 25 | 25 | 25
Completed | 10 | 12 | 18
Not Completed | 15 | 13 | 7
Not completed — Withdrawal by Subject | 9 | 8 | 5
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 5 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | 25mg Meclizine | 50mg Meclizine | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.80 (12.3) | 42.40 (11.60) | 45.80 (10.09) | 43.67 (11.47)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 25 | 75
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 14 | 42
  Male | 12 | 10 | 11 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 14 | 11 | 13 | 38
  White | 11 | 11 | 11 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 25 | 25 | 24 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Change in Expired Air Carbon Monoxide (CO) at End of Week 1
Description: To evaluate the effects of meclizine alone on ad lib smoking, the percent decrease in expired air carbon monoxide (CO) at the end of week 1 (relative to baseline) will be compared (using ANOVA) between each meclizine group and placebo.
Time Frame: After 1 week of treatment (relative to baseline)
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Control | 25mg Meclizine | 50mg Meclizine
Number analyzed (Participants) | 18 | 23 | 25
percentage change | 1.73 (9.03) | -14.11 (5.86) | -.63 (6.85)

2. Primary Outcome: Percentage of Change in Expired Air Carbon Monoxide (CO) at End of Week 3
Description: To evaluate the effects of meclizine as an augmentation treatment in conjunction with nicotine patch, the percent decrease in expired air carbon monoxide (CO) at the end of week 3 (relative to baseline) will be compared (using ANOVA) between each meclizine group and placebo.
Time Frame: After 3 weeks of treatment (relative to baseline)
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Control | 25mg Meclizine | 50mg Meclizine
Number analyzed (Participants) | 18 | 23 | 25
percentage change | -34.05 (11.83) | -54.10 (5.41) | -35.60 (8.72)

3. Secondary Outcome: Number of Participants Completing the Continuous 4 Week Abstinence From Smoking
Description: Continuous 4 week abstinence from smoking (weeks 3-6 post quit date), based on self-reported abstinence confirmed by expired air CO ≤8ppm, will be compared between each meclizine group and placebo, using logistic regression analyses
Time Frame: weeks 3-6 post quit date
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Control | 25mg Meclizine | 50mg Meclizine
Number analyzed (Participants) | 25 | 25 | 25
participants | 2 [.25 to 6.5] | 7 [3.00 to 12.25] | 2 [.25 to 6.5]

4. Secondary Outcome: Percentage of Change of CO at End of Week 1 When Comparing Abstinent Smokers Versus Non-abstinent Smokers
Description: To further validate the association between a decrease in expired air CO before the quit date and subsequent abstinence, the decrease in expired air CO from baseline to week 1 (Session P2) will be compared between abstinent and non-abstinent smokers, using ANOVA.
Time Frame: After 1 week of treatment (relative to baseline)
Population: Abstinent (n=2 "Control", 7 "25mg", 2 "50mg") Non-abstinent (n=16 "Control", 16 "25mg", 23 "50mg")
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Control | 25mg Meclizine | 50mg Meclizine
Number analyzed (Participants) | 18 | 23 | 25
percentage change
  abstinent | 5.00 (15.00) | 2.64 (20.56) | -16.67 (16.67)
  non-abstinent | 1.32 (10.10) | -17.64 (5.66) | -5.37 (7.35)

5. Secondary Outcome: Percentage of Change of CO at End of Week 3 When Comparing Abstinent Smokers Versus Non-abstinent Smokers
Description: To further validate the association between a decrease in expired air CO before the quit date and subsequent abstinence, the decrease in expired air CO from baseline to week 3 (Session P3) will be compared between abstinent and non-abstinent smokers, using ANOVA.
Time Frame: After 3 weeks of treatment (relative to baseline)
Population: Abstinent (n=2 "Control", 7 "25mg", 2 "50mg") Non-abstinent (n=16 "Control", 16 "25mg", 23 "50mg")
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Control | 25mg Meclizine | 50mg Meclizine
Number analyzed (Participants) | 18 | 23 | 25
percentage change
  abstinent | -47.50 (52.50) | -82.77 (10.23) | -56.76 (35.55)
  non-abstinent | -32.13 (12.32) | -47.72 (22.02) | -33.38 (39.74)

ADVERSE EVENTS:
Time Frame: Subjects were receiving study drugs for nine weeks. At each study session during this period subjects completed a questionnaire about side effects. Subjects were also told to contact us between study sessions if side effects were bothersome.
Description: Eight subjects discontinued study participation after the first study session; therefore, no side effects data were collected. Six of these subjects were in the control group, two of these subjects were in the 25mg Meclizine group and none were in the 50mg Meclizine group.
Arm/Group | Control | 25mg Meclizine | 50mg Meclizine
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 14/19 | 14/23 | 15/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=19) | 25mg Meclizine (N=23) | 50mg Meclizine (N=25)
Nausea (Gastrointestinal disorders) | 6 (6) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 2 (2)
Diarrhea / Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Mouth / Throat Irritation (General disorders) | 1 (1) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Coughing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 3 (3)
Irritability (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3)
Difficulty Concentrating (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Drowsiness (Nervous system disorders) | 1 (1) | 5 (5) | 3 (3)
Fatigue (Nervous system disorders) | 2 (2) | 4 (4) | 5 (5)
Nightmares (Nervous system disorders) | 4 (4) | 8 (9) | 3 (3)
Vivid Dreams (Nervous system disorders) | 7 (8) | 12 (12) | 9 (9)
Insomnia (Nervous system disorders) | 5 (6) | 3 (3) | 5 (5)
Itching at Patch Site (Skin and subcutaneous tissue disorders) | 12 (16) | 6 (7) | 7 (7)
Rash at Patch Site (Skin and subcutaneous tissue disorders) | 7 (10) | 3 (3) | 1 (1)
Rash Distant from Patch Site (General disorders) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes